CLINICAL TRIAL: NCT01444183
Title: Pre-emptive Treatment in Epilepsy Using Electronic Diaries: Towards a New Frontier in Epilepsy Therapy
Brief Title: Stress Management Intervention for Living With Epilepsy (SMILE)
Acronym: SMILE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Charles L Shor Foundation for Epilepsy Research (Unknown); University of Cincinnati (Other)
Responsible Party: Principal Investigator, Sheryl Haut, Prof. Dept of Medicine (Critical Care), Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-07-296E
Record Dates: First submitted 2011-09-15; First posted 2011-09-30 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2015-04

CONDITIONS: Epilepsy
Keywords: Epilepsy; seizures; stress reduction
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progressive muscle relaxation (Active Comparator): Subjects practice a progressive muscle relaxation exercise for 15 minutes every AM and 5 minutes every PM
  Interventions: Behavioral: Progressive muscle relaxation
- Sham exercise (Sham Comparator): Subjects practice a sham exercise consisting of focused attention activities
  Interventions: Behavioral: Sham exercise

INTERVENTIONS:
Behavioral: Progressive muscle relaxation — Subjects practice a progressive muscle relaxation exercise for 15 minutes every AM and 5 minutes every PM
  Both groups will practice twice daily, one 15 minute practice in the AM and a 5 minute practice in the PM. An additional 5 minute mid-day practice will occur only when e-diary entries from experience sampling meet specific predetermined criteria.
  Arms: Progressive muscle relaxation
Behavioral: Sham exercise — The focused attention practices will consist of one or more of the following components: movement of body parts, breathing exercises, and writing exercises.
  Both groups will practice twice daily, one 15 minute practice in the AM and a 5 minute practice in the PM. An additional 5 minute mid-day practice will occur only when e-diary entries from experience sampling meet specific predetermined criteria.
  Arms: Sham exercise

SUMMARY:
The study will examine whether a stress reduction intervention reduces the number of seizures in people with drug resistant epilepsy.

DETAILED DESCRIPTION:
The study will examine whether a stress reduction intervention reduces the number of seizures in people with drug resistant epilepsy. In the proposed randomized controlled, double blind trial, the investigators will enroll subjects with frequent seizures, especially those who identify stress as a seizure precipitant. There is an observational phase (8-12 weeks) and a treatment phase (12 weeks). During the observational phase, subjects will be monitored multiple times daily via smart phone devices, in order to identify high risk days for seizures. In the treatment phase, subjects will be randomly assigned to one of two groups receiving different focused attention practices. These behavioral interventions will be administered daily with extra interventions applied on days of higher risk.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above
* English speaking
* Partial epilepsy consistent with ILAE criteria supported by either EEG or MRI data
* Experiencing at least 2 seizures/month
* Reported awareness of all seizures, including seizures in a cluster
* One of the following:

  1. Patient-reported ability to self-predict seizures
  2. Patient-reported awareness of trigger factors, including stress
  3. Patient-reported awareness of premonitory features
* Able to maintain accurate e-diary independently
* Minimum 6th grade reading level as screened by WRAT administration
* Must be on a stable dose of anti-epileptic drugs for at least 30 days prior to study entry
* May be on stable dose of SSRI, SNRI, or atypical antipsychotic for at least 6 months
* May be on a stable dose of benzodiazepines (if so, dose stable for at least 30 days prior to study entry)

For inclusion in clinical trial phase, patient must be/have:

* A minimum of 4 seizures documented in the 8-week baseline phase (or 6 seizures in the 12-week extended baseline phase)
* At least 1 seizure per 4-week period in two of the three 4-week periods in the extended baseline phase
* Diaries satisfactorily completed during baseline phase
* Complied with study requirements during the baseline phase

Exclusion Criteria:

* Non-motor simple partial seizures only
* Concurrent VNS use
* History of suicide attempt within the past 2 years
* Current suicidality
* Not competent to sign consent
* Status epilepticus within the previous 6 months
* Began regularly using behavioral techniques for stress reduction within past 3 months
* Did not benefit from an adequate trial of a valid stress reduction technique
* Progressive neurologic condition that the investigator believes would affect seizure frequency
* Any history of substance abuse within the previous 2 years
* History of poor medication compliance as judged by the investigator
* Psychiatric illness that requires change in medication dose
* Any medical or psychiatric condition that would impair reliable participation in the trial
* Intermittent use of benzodiazepines (if used for sleep, will be determined case by case)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2012-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in seizure frequency | End of baseline and end of 12 week clinical trial

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl Haut, MD, Principal Investigator — Montefiore Medical Center; Michael Privitera, MD, Principal Investigator — University of Cincinnati; Susannah Cornes, MD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California San Francisco, San Francisco, California
  - Montefiore Medical Center, The Bronx, New York
  - University of Cincinnati, Cincinnati, Ohio

REFERENCES:
- [Background] Hall CB, Lipton RB, Tennen H, Haut SR. Early follow-up data from seizure diaries can be used to predict subsequent seizures in same cohort by borrowing strength across participants. Epilepsy Behav. 2009 Mar;14(3):472-5. doi: 10.1016/j.yebeh.2008.12.011. Epub 2009 Jan 10. PMID 19138755
- [Background] Haut SR, Hall CB, Masur J, Lipton RB. Seizure occurrence: precipitants and prediction. Neurology. 2007 Nov 13;69(20):1905-10. doi: 10.1212/01.wnl.0000278112.48285.84. PMID 17998482
- [Background] Heron KE, Smyth JM. Ecological momentary interventions: incorporating mobile technology into psychosocial and health behaviour treatments. Br J Health Psychol. 2010 Feb;15(Pt 1):1-39. doi: 10.1348/135910709X466063. Epub 2009 Jul 28. PMID 19646331
- [Background] Nickel C, Kettler C, Muehlbacher M, Lahmann C, Tritt K, Fartacek R, Bachler E, Rother N, Egger C, Rother WK, Loew TH, Nickel MK. Effect of progressive muscle relaxation in adolescent female bronchial asthma patients: a randomized, double-blind, controlled study. J Psychosom Res. 2005 Dec;59(6):393-8. doi: 10.1016/j.jpsychores.2005.04.008. PMID 16310021
- [Derived] Privitera M, Haut SR, Lipton RB, McGinley JS, Cornes S. Seizure self-prediction in a randomized controlled trial of stress management. Neurology. 2019 Nov 26;93(22):e2021-e2031. doi: 10.1212/WNL.0000000000008539. Epub 2019 Oct 23. PMID 31645468
- [Derived] Haut SR, Lipton RB, Cornes S, Dwivedi AK, Wasson R, Cotton S, Strawn JR, Privitera M. Behavioral interventions as a treatment for epilepsy: A multicenter randomized controlled trial. Neurology. 2018 Mar 13;90(11):e963-e970. doi: 10.1212/WNL.0000000000005109. Epub 2018 Feb 14. PMID 29444968